CLINICAL TRIAL: NCT06709495
Title: Phase 1/2 Trial to Evaluate the Safety and Efficacy of PEEL-224 in Combination With Vincristine and Temozolomide in Adolescents and Young Adults With Relapsed or Refractory Sarcomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David S Shulman, MD (Other)
Collaborators: Peel Therapeutics Inc (Industry)
Responsible Party: Sponsor-Investigator, David S Shulman, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-591
Record Dates: First submitted 2024-11-17; First posted 2024-11-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma; Sarcoma, Ewing; Desmoplastic Small Round Cell Tumor; Refractory Sarcoma; Osteosarcoma; Rhabdomyosarcoma
Keywords: Sarcoma; Sarcoma, Ewing; Desmoplastic Small Round Cell Tumor; Refractory Sarcoma; Relapsed Sarcoma; osteosarcoma; rhabdomyosarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Ewing; Desmoplastic Small Round Cell Tumor; Osteosarcoma; Rhabdomyosarcoma | interventions — Temozolomide; Vincristine; pegfilgrastim; Filgrastim; Granulocyte Colony-Stimulating Factor; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Phase 1: Dose Escalation PEEL-224 Dose Level 0 (Experimental): Up to 15 participants will be enrolled using a Bayesian design, the Continual Reassessment Method (CRM), to determine the maximum tolerated dose of PEEL-224 and starting at Dose Level 0. Transition to a lower dose level will be determined by types of dose-limiting toxicities observed per the protocol.
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 1: Dose Escalation PEEL-224 Dose Level -1A (Experimental): Transition to a lower dose level will be determined by types of dose-limiting toxicities observed per the protocol, otherwise establishment of the MTD/RP2D will be according to the CRM model.
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 1: Dose Escalation PEEL-224 Dose Level -1B (Experimental): Transition to a lower dose level will be determined by types of dose-limiting toxicities observed per the protocol, otherwise establishment of the MTD/RP2D will be according to the CRM model.
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 1: Dose Escalation PEEL-224 Dose Level -2 (Experimental): Establishment of the MTD/RP2D will be according to the CRM design.
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 1: Dose Escalation PEEL-224 Dose Level 1 (Experimental): Escalation to Dose Level 2 or establishment of the MTD/RP2D will be determined by the CRM design.
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 1: Dose Escalation PEEL-224 Dose Level 2 (Experimental): Establishment of the MTD/RP2D will be determined by the CRM design.
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 2: Dose Expansion Ewing Sarcoma (Experimental): Administration of PEEL-224 will be at the RP2D, and safety monitoring rules will be applied for the occurrence of dose-limiting toxicities. 15 participants will be enrolled and will complete:
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 2: Dose Expansion DSRCT (Experimental): Administration of PEEL-224 will be at the RP2D, and safety monitoring rules will be applied for the occurrence of dose-limiting toxicities. 15 participants will be enrolled and will complete:
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim
- Phase 2: Dose Expansion Other Sarcoma (Experimental): Administration of PEEL-224 will be at the RP2D, and safety monitoring rules will be applied for the occurrence of dose-limiting toxicities. 15 participants will be enrolled and will complete:
  * Baseline visit with assessments and imaging
  * Cycle 1 (21 day cycle):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
    * Day 10: Myeloid growth factor (Pegfilgrastim or Filgrastim) administration 1x daily
  * Cycle 2 through End of Treatment (21 day cycles):
    * Days 1 through 5: Predetermined dose of Temozolomide 1x daily
    * Days 1 and 8: Predetermined dose of PEEL-224 1x daily and predetermined dose of Vincristine 1x daily
  * Imaging every 2 cycles until Cycle 6 and then every 3 cycles
  * End of study visit
  Interventions: Drug: PEEL-224; Drug: Temozolomide; Drug: Vincristine; Biological: Pegfilgrastim; Biological: Filgrastim

INTERVENTIONS:
Drug: PEEL-224 — Topoisomerase 1 inhibitor, 200mg amber vial, via intravenous (into the vein) infusion per protocol.
Drug: Temozolomide — Alkylating agent, 5, 20, 100, 140, 180, or 250 mg capsule, taken orally per standard of care.
  Other Names: Temodar; Temodal
Drug: Vincristine — Vinca alkaloid, 1 or 2mL vials, via intravenous (into the vein) infusion per institutional policy.
Biological: Pegfilgrastim — Myeloid growth factor administered per institutional standards.
  Other Names: Neupogen
Biological: Filgrastim — Myeloid growth factor administered per institutional standards.
  Other Names: Nivestym; Granix; Zarxio; Filgrastim-Aafi; Filgrastim-Sndz; Tbo-Filgrastim,; RHG-CSF

SUMMARY:
This research is being done to test a new drug called PEEL-224 in combination with two commercially available drugs, Vincristine and Temozolomide, and to determine how effective this combination of drugs is at treating Ewing Sarcoma (EWS) and Desmoplastic Small Round Cell Tumor (DSRCT), as well as multiple other kinds of sarcomas.

The names of the study drugs and biological agents involved in this study are:

* PEEL-224 (a type of Topoisomerase 1 inhibitor)
* Vincristine (A type of vinca alkaloid)
* Temozolomide (A type of alkylating agent)
* Pegfilgrastim or Filgrastim (types of Myeloid growth factors)

DETAILED DESCRIPTION:
This is an open-label, single-arm, non-randomized, phase I/II trial to test a new drug called PEEL-224 in combination with two commercially available drugs, Vincristine and Temozolomide, and to determine how effective this combination of drugs is at treating Ewing Sarcoma (EWS) and Desmoplastic Small Round Cell Tumor (DSRCT), as well as multiple other kinds of sarcomas. This is the first time that PEEL-224 will be given in combination with Vincristine and Temozolomide to humans.

In Phase 1, the safety and tolerability of PEEL-224 in combination with Vincristine and Temozolomide will be assessed by dose escalation and establishment of a Recommended Phase 2 Dose. In Phase 2 the efficacy of the drug combination will be assessed in three separate cohorts of participants.

The U.S. Food and Drug Administration (FDA) has not approved PEEL-224 as a treatment for Relapsed or Refractory Sarcoma.

The U.S. Food and Drug Administration (FDA) has not approved Vincristine and Temozolomide for Relapsed or Refractory Sarcoma, but it has been approved for other uses.

The research study procedures include screening for eligibility, study treatment in-clinic visits, X-rays, Computerized Tomography (CT) scans, Magnetic Resonance Imaging (MRI) scans, or Positron Emission Tomography (PET) scans, blood tests, urine tests, and electrocardiograms (ECGs).

Participants will receive study treatment for up to 34 cycles (approximately 2 years) and will be followed for up to 1 year after the last participant has received the last dose of treatment.

It is expected that about 63 people will take part in this research study.

PEEL Therapeutics is funding this research study by providing the study drug, PEEL-224.

ELIGIBILITY:
Inclusion Criteria:

-Patients in all cohorts must have relapsed or refractory disease after standard therapy.

Inclusion Criteria Phase 1 (only) diagnosis requirements:

-Patients must have:

* Evaluable or measurable disease; and
* Histologic diagnosis of sarcoma

Inclusion Criteria Phase 2 (only) diagnosis requirements

* EWS cohort: Patients must have:

  * RECIST measurable disease at study entry;
  * Histologic diagnosis consistent with Ewing sarcoma; and
  * Molecular evidence of a FET-ETS family translocation including but not limited to any of the following:

    * EWSR1::FLI1, EWSR1::ERG, EWSR1::ETV1, EWSR1::ETV4, EWSR1::FEV, FUS::FLI1, FUS::ERG
* DSRCT cohort: Patients must have:

  * RECIST measurable disease at study entry;
  * Histologic diagnosis consistent with DSRCT; and
  * Molecular evidence of an EWSR1::WT1 fusion
* Other sarcoma cohort: Patients must have:

  * RECIST evaluable or measurable disease; and
  * Histologic diagnosis of sarcoma. Patients with EWS or DSRCT with evaluable but not measurable disease may participate in this cohort.
  * Slots in this cohort will include three dedicated slots for patients with rhabdomyosarcoma, three dedicated slots for patients with osteosarcoma and three dedicated slots for patients with other translocation-associated round cell sarcomas.
* Age: ≥ 12 years and ≤ 49 years.
* Weight: Patients must be ≥ 40 kg.
* Performance Status: Karnofsky ≥ 50% for patients >16 year of age and Lansky ≥ 50% for patients ≤ 16 years of age. (see Appendix A for definitions of Lansky and Karnofsky Performance Status).
* Participants must meet the following organ and marrow function as defined below: Adequate Bone Marrow Function:

  * Hematologic Requirements for Subjects without Bone Marrow Involvement by

Disease:

* Absolute neutrophil count (ANC) ≥ 1,000/uL
* Platelet count ≥100,000/uL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)

  --Hematologic Requirements for Subjects with Bone Marrow Involvement by Disease:
* ANC ≥750 /uL
* Platelets ≥50,000 /uL (may receive platelet transfusions) Not known to be refractory to red cell and/or platelet transfusions.

  --Adequate Renal Function: Creatinine clearance or radioisotope GFR ≥70ml/min/1.73 m2 or A serum creatinine based on age/sex as follows:
* Age: 12 to < 13 years, Maximum Serum Creatinine (mg/dL): Male 1.2, Female 1.2
* Age 13 to < 16 years, Maximum Serum Creatinine (mg/dL): Male 1.5, Female 1.4

  ---≥ 16 years, Maximum Serum Creatinine (mg/dL): Male 1.7, Female 1.4

  --Adequate Liver Function:
* Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age
* SGPT (ALT) ≤110 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.

  * Adequate Cardiac Function: QTc < 480 msec

    -Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy except organ function as noted above. Patients must meet the following minimum washout periods prior to enrollment:
  * Myelosuppressive chemotherapy: At least 14 days after the last dose of myelosuppressive chemotherapy
  * Radiotherapy:
* At least 14 days after local XRT (small port, including cranial radiation);
* At least 90 days must have elapsed after prior TBI, craniospinal XRT or if >50% radiation of pelvis;
* At least 42 days must have elapsed if other substantial BM radiation.

  * Small molecule biologic therapy: At least 7 days following the last dose of a biologic agent.
  * Monoclonal antibody: At least 21 days must have elapsed after the last dose of antibody.
  * Myeloid and platelet growth factors: At least 14 days following the last dose of long-acting myeloid growth factor (e.g. Neulasta) or 7 days following short-acting myeloid or platelet growth factor.
  * Autologous hematopoietic stem cell transplant and stem cell boost: Patients must be at least 60 days from day 0 of an autologous stem cell transplant or stem cell boost.
  * Cellular Therapies (e.g., CART, NK-cell based therapy): The patient must be and at least 42 days from cellular therapy administration.
  * Major Surgery: At least 2 weeks from prior major surgical procedure. Note: Biopsy, CNS shunt placement/revision, and central line placement/removal are not considered major.
  * Irinotecan, liposomal irinotecan, and/or temozolomide: Patients may have received prior irinotecan, liposomal irinotecan, and/or temozolomide. NOTE: Patients who have had progressive disease while receiving irinotecan and temozolomide in combination will be excluded from the Phase 2 EWS and DSRCT cohorts only.

    -For patients with metastatic disease to the CNS enrolling to the phase 1 portion of the trial or the "other sarcoma" cohort, any baseline neurologic deficits (including seizure) must be stable for at least one week prior to study enrollment. Patients with CNS metastatic disease receiving corticosteroids must be on a stable or decreasing dose at time of study entry.
  * Patients with CNS metastatic disease will not be eligible for the phase 2 EWS and DSRCT cohorts.

    * Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
    * The effects of PEEL-224 in combination with temozolomide and vincristine on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of PEEL-224 administration.
    * Ability to understand and/or the willingness of the patient (or parent or legally authorized representative, if minor) to provide informed consent, using an institutionally approved informed consent procedure.
    * Any participant must obtain prior approval from insurance to reimburse oral temozolomide for the duration of the study or agree to self-pay for oral temozolomide.

Exclusion Criteria:

* Patients who have received prior treatment with PEEL-224.
* Patients who have had progressive disease while receiving irinotecan and temozolomide in combination will be excluded from the Phase 2 EWS and DSRCT cohorts only.
* Participants who are receiving any other anti-cancer agents for this condition.
* Patients receiving strong P450 CYP1A2 and CYP3A4 inhibitors and/or inducers with 14 days of the first planned dose of PEEL-224. NOTE: levofloxacin is permitted and preferred over ciprofloxacin for patients needing a fluoroquinolone.
* Patients who have received a solid organ or allogeneic stem cell transplant
* Pregnant participants, given that the effects of PEEL-224 on the developing human fetus are unknown.
* Breastfeeding mothers, because there is an unknown risk for adverse events in nursing infants secondary to treatment of the mother with PEEL-224.
* Patients with a history of allergic reactions attributed to PEGylated drugs, camptothecins, temozolomide or vincristine.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 12 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) (Phase 1) | Up to 35 days
  The MTD is determined by a Continual Reassessment Method (CRM) design and defined as the dose level with the posterior probability of dose-limiting toxicity (DLT) closest to the target toxicity rate of 0.3 with a maximum sample size of 15. The DLT observation period is up to 35 days long, beginning at the first dose of any of the three drugs in cycle 1 and ending at the occurrence of a DLT.
Number of Participants with Dose-Limiting Toxicities (Phase 1) | Up to 35 days
  Any ≥ Grade 2 CTCAE v5 adverse events that are possibly, probably, or definitely attributable to the combination of Vincristine, PEEL-224, and Temozolomide and within the first 35 days, beginning at the first dose of any of the three drugs in cycle 1 and ending at the occurrence of DLT or at the start of treatment in cycle 2 (whichever occurs first). To be evaluable for dose-limiting toxicity, a participant must also receive at least 75% of prescribed agents in cycle 1 and be followed for at least 35 days during cycle 1 or to the start of cycle 2 (whichever occurs first).
Number of Participants with DLTs (Phase 2) | Up to 35 days
  A safety monitoring rule will be applied to Phase 2 of the study for the overall participant cohort. The DLT observation period is up to 35 days long, beginning at the first dose of any of the three drugs in cycle 1 and ending at the occurrence of DLT or at the start of treatment in cycle 2 (whichever occurs first).
Objective Response Rate EWS Cohort (Phase 2) | Up to 5 years (based on accrual duration of 2 years)
  ORR is defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Evaluable participants must have measurable disease at screening, be treated at RP2D dose, have received at least one dose of study drug, and either have evidence of clinical progression or have had at least one follow-up disease evaluation of their RECIST measurable disease after initiation of protocol therapy. The proportion of responders is calculated as the (number of responders) / (number of evaluable participants).
Objective Response Rate DSRCT Cohort (Phase 2) | Up to 5 years (based on accrual duration of 2 years)
  ORR is defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Evaluable participants must have measurable disease at screening, be treated at RP2D dose, have received at least one dose of study drug, and either have evidence of clinical progression or have had at least one follow-up disease evaluation of their RECIST measurable disease after initiation of protocol therapy. The proportion of responders is calculated as the (number of responders) / (number of evaluable participants).

SECONDARY OUTCOMES:
Objective Response Rate Other Sarcoma Cohort | Up to 5 years (based on accrual duration of 2 years)
  ORR is defined as the percentage of participants achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Evaluable participants must have measurable disease at screening, be treated at RP2D dose, have received at least one dose of study drug, and either have evidence of clinical progression or have had at least one follow-up disease evaluation of their RECIST measurable disease after initiation of protocol therapy. The proportion of responders is calculated as the (number of responders) / (number of evaluable participants).
Median Progression-Free Survival (PFS) Other Sarcoma Cohort | Approximately 2 years
  Progression-Free Survival (PFS) based on the Kaplan-Meier method is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Overall Survival (OS) Other Sarcoma Cohort | Up to 5 years (based on accrual duration of 2 years)
  Overall Survival (OS) based on the Kaplan-Meier method is defined as the time from registration to death due to any cause, or censored at date last known alive.
Median PFS EWS Cohort | Approximately 2 years
  PFS based on the Kaplan-Meier method is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
OS EWS Cohort | Up to 5 years (based on accrual duration of 2 years)
  OS based on the Kaplan-Meier method is defined as the time from registration to death due to any cause, or censored at date last known alive.
Median PFS DSRCT Cohort | Approximately 2 years
  PFS based on the Kaplan-Meier method is defined as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
OS DSRCT Cohort | Up to 5 years (based on accrual duration of 2 years)
  OS based on the Kaplan-Meier method is defined as the time from registration to death due to any cause, or censored at date last known alive.
Peak Plasma Concentration (Cmax) of PEEL-224 | Days 1, 2, 3, and 8 of Cycle 1 (21 days per cycle)
  Cmax will be estimated within the cohort of evaluable participants 12 years and older who received PEEL-224 given on a 2-week on and 1-week off schedule.
Area Under the Plasma Concentration Versus Time Curve (AUC) of PEEL-224 | Days 1, 2, 3, and 8 of Cycle 1 (21 days per cycle)
  AUC will be estimated within the cohort of evaluable participants 12 years and older who received PEEL-224 given on a 2-week on and 1-week off schedule.
Peak Time (Tmax) of PEEL-224 | Days 1, 2, 3, and 8 of Cycle 1 (21 days per cycle)
  Tmax will be estimated within the cohort of evaluable participants 12 years and older who received PEEL-224 given on a 2-week on and 1-week off schedule.
Circulating Tumor DNA (ctDNA) Burden EWS Cohort at Baseline | Baseline
  ctDNA burden is the amount of circulating tumor DNA (ctDNA) present in the bloodstream, reflecting the extent of tumor-derived DNA shed into circulation. A next generation sequencing or PCR-based approach will be used to detect ctDNA.
ctDNA Burden EWS Cohort at Day 8 | Day 8
  ctDNA burden is the amount of circulating tumor DNA (ctDNA) present in the bloodstream, reflecting the extent of tumor-derived DNA shed into circulation. A next generation sequencing or PCR-based approach will be used to detect ctDNA.
ctDNA Burden DSRCT Cohort at Baseline | Baseline
  ctDNA burden is the amount of circulating tumor DNA (ctDNA) present in the bloodstream, reflecting the extent of tumor-derived DNA shed into circulation. A next generation sequencing or PCR-based approach will be used to detect ctDNA.
ctDNA Burden DSRCT Cohort at Day 8 | Day 8
  ctDNA burden is the amount of circulating tumor DNA (ctDNA) present in the bloodstream, reflecting the extent of tumor-derived DNA shed into circulation. A next generation sequencing or PCR-based approach will be used to detect ctDNA.
≥ Grade 2 Treatment-Related Toxicity Rate (Phase 1) | Approximately 2 years
  The percentage of participants that experience a maximum grade 2-5 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms. From start of protocol therapy until 30 days after last dose of temozolomide, vincristine or PEEL-224, which ever occurs last.
≥ Grade 2 Treatment-Related Toxicity Rate (Phase 2) | Approximately 2 years
  The percentage of participants who experience ≥ Grade 2 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms. From start of protocol therapy until 30 days after last dose of temozolomide, vincristine or PEEL-224, which ever occurs last.
Median Duration of Overall Response (DOR) (Phase 2) | Approximately 2 years
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation)
Median Duration of Complete Response (CR) (Phase 2) | Approximately 2 years
  The duration of CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented, or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Median Duration of Stable Disease (Phase 2) | Approximately 2 years
  Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.

CONTACTS AND LOCATIONS:
Overall Officials: David Shulman, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu